CLINICAL TRIAL: NCT05368454
Title: Randomized Controlled Trial to Evaluate the Efficacy of an Integrated Lifestyle Management Solution With Continuous Glucose Monitoring for Type 2 Diabetes
Brief Title: Evaluation of a Digital Diabetes Self-Management Education and Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omada Health, Inc. (Industry)
Collaborators: Abbott Diabetes Care (Industry); Evidation Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022 V 5.0
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Solution (Experimental)
  Interventions: Behavioral: Online Diabetes Self-Management Education and Support (DSMES) Program
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Online Diabetes Self-Management Education and Support (DSMES) Program — An online program for Diabetes Self-Management, Education and Support (DSMES) that includes personal coaching by a certified Diabetes Care and Education Specialist (CDCES), tracking tools, and FreeStyle Libre CGMs, a wearable sensor with data scanning ability accessed through the smartphone app.
  Arms: Integrated Solution
Behavioral: Standard of Care — All participants randomized to the standard of care/control arm will be asked to continue with their current care plan and care team for management of their diabetes.
  Arms: Standard of Care

SUMMARY:
The goal of this study is to examine the efficacy of an integrated solution, defined as a combination of the Abbott FreeStyle Libre 14-day CGM sensor and the Omada care team's receipt of real-time, continuous glucose data from the sensor and incorporation of this data into their care delivery within the context of the Omada for Diabetes program for adults with Type 2 Diabetes (T2D). This randomized control trial will test the impact of the integrated solution on HbA1c, CGM-derived metrics and other relevant diabetes management outcomes over six months compared to the current standard of care.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) contributes substantially to morbidity and mortality in the US. Lifestyle management is a fundamental component of care for T2D. This includes self-management education and support, medical nutrition therapy, physical activity, smoking cessation counseling, and psychosocial care for the person with diabetes. Diabetes self-management education and support (DSMES) specifically pertains to helping people acquire the knowledge, skills, and ability for diabetes self-care, and assisting people to engage in the health-related behaviors needed to manage this condition on an ongoing basis. Research has shown that DSMES programs that target behavioral changes with intensive counseling and support lead to improved glucose control.

In recent years, technology-enabled platforms have been developed to deliver self-management support and education virtually, and commercial products are common. These platforms allow people with chronic diseases to access self-management support and education through their personal mobile devices (e.g., smartphones, tablets, laptops) and eliminate the need to travel to physical facilities for diabetes education sessions. The increased convenience brings potential to increase access, availability, and acceptability.

The development of Continuous Glucose Monitoring (CGM) has further advanced care and management of T2D. In particular, real-time CGM allows the person to view real-time glucose readings and patterns over time, without the need for painful finger sticks. While the majority of studies of CGM have been conducted with people with T2Ds using insulin, some clinical trials have shown that the use of real-time CGM is associated with improvements in glycemic control in people with T2D not using insulin.

The current standards of care for diabetes recommend CGM use for people with Type 1 and 2 diabetes when it is coupled with "robust diabetes education, training and support". However, there is a lack of well-integrated solutions that combine the potential benefit of both digitally delivered DSMES and CGM in a seamless way. Therefore, the purpose of this study is to examine the efficacy of a novel integrated solution of a digitally delivered T2D self-management education and support program with a continuous glucose monitor (CGM) built into the digital platform. The randomized control trial will test the impact of the novel solution for improving HbA1c and related CGM-derived outcomes and relevant diabetes management outcomes over six months related to the current standard of care.

ELIGIBILITY:
INCLUSION CRITERIA

1. 18 years or older
2. Lives in the United States and has a valid mailing address
3. Speaks, reads, and understands English as the primary language
4. Be willing and able to provide written, signed, and dated informed consent
5. Has a self-reported diagnosis of type 2 diabetes prior to enrollment for at least 6 months
6. Self-reports HbA1c value ≥8.0% from most recent test taken within the past 6 months
7. Treatment regimen includes diet and exercise alone, oral glucose lowering medication, non-insulin injectable medications, basal insulin and/or combination of basal insulin plus oral medications. No more than 15% of the total sample may be on combination basal insulin/oral medication.

   a. If the regimen is basal insulin with oral medications, the participant must have initiated basal insulin in addition to oral medication at least 6 months prior to enrollment.
8. Currently on medication regimen for at least 3 months prior to enrollment
9. HbA1c greater than or equal to 8.0% as demonstrated by laboratory HbA1c at secondary screening
10. Has a compatible smartphone running either Android OS 5.0 or higher, or iPhone 7 or later, running iOS 11 or higher with an on-going data plan
11. Is willing to set up an online account using the Omada Health Program/app and LibreLink app, and agree to share their CGM data with designated health care providers connected to the study.
12. Must be willing to complete all study tasks as specified by the protocol
13. Must report being compliant with their diabetes management plan and must be willing to adhere to their medication regimen throughout the study.
14. Not currently in another clinical trial

EXCLUSION CRITERIA

1. Type 1 diabetes or a history of diabetic ketoacidosis
2. Self-reported HbA1c < 8.0% or does not know their HbA1c level
3. Self-reported condition leading to life expectancy < 12 months
4. Pregnant, is attempting to conceive or is not willing and able to practice birth control during the study duration (applicable to female participants who are able to become pregnant only)
5. Currently has self-reported skin lesions, scarring, redness, infection or edema at the application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. This includes known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin
6. Has X-ray, MRI or CT appointment scheduled during the study periods of CGM measurement with the FreeStyle Libre Pro, and the appointment(s) cannot be rescheduled
7. Currently using mealtime bolus injections of insulin, premixed insulin formulations or a continuous subcutaneous infusion of insulin
8. Visual impairment that would prohibit ability to view sensor data or use the Omada platform
9. Has had any of the following in the past 3 months:

   * Transient ischemic attack or stroke
   * Heart attack (myocardial infarction)
   * Hospitalization for congestive heart failure
   * Cardiac surgery (such as coronary artery bypass grafting (CABG), coronary artery stenting)
   * If it has been > 3 months since any of the above, applicant must be medically cleared by their primary physician to exercise
10. Bariatric/gastric bypass surgery, including gastric sleeve, gastric balloon within the past 6 months
11. Participation in other research studies involving medication or device within 1 month prior to enrollment
12. Organ transplant (kidney, liver, etc.) within the past 6 months
13. Recent (within the last 6 months) or planned cancer treatment (chemotherapy, radiation, bone marrow transplant, cancer-related surgery - not including hormonal chemotherapy, such as tamoxifen)
14. Self-reported renal impairment, defined as estimated glomerular filtration rate <30 mL/min/1.73 m2
15. Language barriers precluding comprehension of study activities and informed consent 16. Currently on a routine regimen of glucocorticoids or psychotropic medications 17. Self-reported alcohol or substance abuse issue or dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 3 months, 6 months
  Non-fasting venous blood sample

SECONDARY OUTCOMES:
Change in daily Time in Range [70-180] mg/dL | Baseline, 3 months, 6 months
  Derived from continuous glucose monitor
Change in body weight | Baseline, 3 months, 6 months
  Measured with a digital weight scale in stocking feet
Change in resting blood pressure | Baseline, 3 months, 6 months
  Collected with an automated, calibrated blood pressure monitor with self-inflating cuff
Change in diabetes distress | Baseline, 3 months, 6 months
  The Diabetes Distress Scale, a 17-item self-report questionnaire, that captures four dimensions: emotional burden, regimen distress, interpersonal distress and physician distress related to diabetes and diabetes self-care

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Linke, PhD, Study Director — Omada Health, Inc.; David Kerr, MBChB, DM, FRCPE, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No